CLINICAL TRIAL: NCT03554707
Title: A Pilot Study of SGT-53 in Conjunction With Irradiation and Chemotherapy in Children With Recurrent or Progressive CNS Malignancies
Brief Title: SGT-53 in Children With Recurrent or Progressive CNS Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SynerGene Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGT53-00-1
Record Dates: First submitted 2018-05-17; First posted 2018-06-13 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Childhood CNS Tumor
Keywords: Childhood CNS tumor; Recurrent CNS malignancies; Progressive CNS malignancies; Refractory CNS malignancies
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Radiation; Irinotecan; irinotecan sucrosofate; Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SGT-53 with radiation or drugs (Experimental): Radiation phase: SGT-53 will be given at 2.1 mg DNA/m2 twice weekly for the first week of radiation therapy, and then increase to 2.8 mg DNA/m2 twice weekly. Radiation therapy will be administered as per clinical care, with a target of fifteen (15) fractions, but patients with other clinically-determined radiation plans will be allowed.
  Chemotherapy phase: SGT-53 will be administered at the highest tolerated dose given during radiation phase. Irinotecan will be given at a dose of 50mg/m2/dose IV daily for five days in a 4-week cycle. Temozolomide will be given at a dose of 100mg/m2 PO daily for five days in a 4-week cycle and bevacizumab will be given at a dose of 10mg/kg IV every two weeks in a 4-week cycle.
  Interventions: Genetic: SGT-53; Radiation: Radiation; Drug: Irinotecan; Drug: Temozolomide; Drug: Bevacizumab

INTERVENTIONS:
Genetic: SGT-53 — 2.1 mg DNA/m2 or 2.8 mg DNA/m2 twice weekly
Radiation: Radiation — Standard radiation plan
Drug: Irinotecan — 50mg/m2/dose IV daily for five days in a 4-week cycle
  Other Names: Camptosar; Onivyde
Drug: Temozolomide — 100mg/m2 PO daily for five days in a 4-week cycle
  Other Names: Temodar
Drug: Bevacizumab — 10mg/kg IV every two weeks in a 4-week cycle
  Other Names: Avastin

SUMMARY:
An early phase 1 for pediatric patients with recurrent or progressive CNS malignancies

DETAILED DESCRIPTION:
This clinical trial is a early phase 1, open label, single center, single arm study of the combination of intravenously administered SGT-53 and irradiation and/or chemotherapy in pediatric patients with recurrent or progressive CNS malignancies. The objective of the study is to establish the safety and feasibility of administration of SGT-53 in conjunction with conventional radiotherapy and/or chemotherapy in children with recurrent or refractory CNS malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a recurrent, progressive, or refractory CNS malignancy for which there are not known curative options. Low-grade glioma, craniopharyngioma, and other non-malignant CNS tumors are excluded.
* Tumor must be measureable, defined as a tumor that can be accurately measured in two perpendicular dimensions on MRI.
* Patients with metastatic disease are eligible but must have at least one target lesions which is measurable.
* Patients must have available archival (formalin-fixed paraffin embedded) or fresh tumor tissue for correlative studies.
* Patients must be >1yrs and <21 years of age.
* Must have recovered from all surgical interventions prior to the start of the Radiation and Chemotherapy Phases.
* Patients must have recovered from the acute effects of prior therapy.
* There is a maximum of 3 previous myelosuppressive therapy regimens. However, there is no maximum number of therapeutic courses.
* Patients must have received their last dose of known myelosuppressive therapy at least three (3) weeks prior to receipt of SGT-53.
* Patients must have received their last dose of biological agent >7 days prior to receipt of SGT-53.
* Patients must be far enough from previous irradiation that in the opinion of a radiation oncologist using standard fractionation is deemed to be reasonable from a clinical standard of care perspective.
* Patients who are receiving dexamethasone or other corticosteroids must be on a stable or decreasing dose for at least one (1) week prior to enrollment.
* Patients must have received their last dose of any short acting growth factor at least one week prior to treatment, for long acting or pegylated growth factors, the last dose must be at least two (2) weeks prior to start of treatment.
* Patients with neurologic deficits must have deficits that have been stable in grade for a minimum of one week prior to enrollment.
* Performance status (Karnofsky PS for >16yrs, or Lansky PS for <16yrs) assessed within two weeks must be >50.
* Patients must have normal organ and marrow function.
* All patients of childbearing or child fathering potential must be willing to use an acceptable form of birth control while being treated on this study.
* Female patients must not be pregnant or nursing. Female patients must also have a negative serum pregnancy test at the time of enrollment.
* Patient and/or guardian have the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria:

* Patients with any clinically significant unrelated systemic illness (serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that is likely to interfere with ability to tolerate study therapy or study procedure results.
* Patients with low-grade gliomas, craniopharyngioma, or extracranial tumors with CNS metastases.
* Patients who are receiving any other investigational drug therapy.
* Patients who require therapeutic anti-coagulation.
* Patients who in the opinion of the investigator cannot adhere to protocol requirements.
* Patients with history of clinically significant clot or hemorrhage are eligible but will not receive bevacizumab during chemotherapy regimen.
* Unavailability of the chemotherapy due to insurance coverage or other logistical issues is an ineligibility criterion.
* Patients may not be on immunosuppressive therapy, including corticosteroids (with the exception of physiologic replacement, defined as 0.75mg/m2/day) at time of enrollment. However, patients who require intermittent use of bronchodilators or local steroid injections will not be excluded from the study.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | up to 13 months
  An adverse event (AE) was any untoward medical occurrence that began or worsened in grade after the start of study drug through 30 days after the last dose. The safety will be assessed by the number and severity of any AE or serious adverse events (SAE) experienced by the patients, and by their relationship to the study drug SGT-53 (e.g. definitely, probably, possibly, unlikely or unrelated). Severity will be graded according to NCI CTCAE version 4.0.

SECONDARY OUTCOMES:
Response Rate | 36 months
  The response rate will be calculated from the percentage of patients whose cancer shrinks or disappears after treatment.
Duration of Response | 36 months
  The duration of response will be the time calculated from documentation of tumor response as indicated by response criteria, to disease progression.
Overall Survival | 36 months
  Overall survival will be calculated from date of original diagnoses to death and also from the date of study registration to death.
Progressive-Free Survival (PFS) | 36 months
  PFS will be calculated at all times during follow-up, with particular interest in the 6-month time point. Progression free survival will be calculated from date of first treatment to the date of first observation of progressive disease, non-reversible neurological progression or increasing steroid requirements (applies to stable disease only), death due to any cause, or early discontinuation of treatment.
Characterization of Phenotype of Patients | 4-5 days
  Tissue will be obtained from each enrolling patient for subsequent testing for TP53 pathway functionality, including assessment of mdm2, p21, and other mutation or expression alterations. This analysis will also include measures of commonly assessed polymorphisms, including MGMT methylation assessment, ATRX mutation among others.
Feasibility of Droplet PCR Assays to Monitor for Tumor Burden | 12 months
  Droplet PCR will be used to assess for the presence of circulating tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Hwang, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided